CLINICAL TRIAL: NCT05607290
Title: Clinical Course of Alcohol Use Disorder Recovery
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Florida (Other)
Responsible Party: Principal Investigator, Robert Schlauch, Principal Investigator, University of South Florida
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1R01AA030005-01A1 (NIH)
Record Dates: First submitted 2022-10-17; First posted 2022-11-07 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Alcohol Use Disorder
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Other): Empirical supported psychotherapy for alcohol use disorder (Cognitive-Behavioral Therapy, Motivational Interviewing).
  Interventions: Behavioral: Cognitive-Behavioral Treatment

INTERVENTIONS:
Behavioral: Cognitive-Behavioral Treatment — 12 sessions of Cognitive-Behavioral Treatment for Alcohol Use Disorder

SUMMARY:
The goal of this single-arm clinical trial is to better understand the ways in which individuals seeking treatment recover from Alcohol Use Disorder (AUD). The main aims are to:

* To establish operational definitions of types of change in relation to National Institute on Alcohol Abuse and Alcoholism's (NIAAA) new definition of recovery, and to distinguish between treatment response, remission versus recovery, and relapse versus recurrence.
* To describe patterns of recovery, including the frequency of within-person transitions between types of change in clinical course to better understand the dynamic nature of recovery.
* To examine the predictive relationships between theoretically important cognitive, behavioral, and affective process variables and changes during recovery, with a focus on how people initiate versus maintain change.

Participants will:

* Receive 12 weeks of psychotherapy for Alcohol Use Disorder
* Complete brief assessments after each treatment session.
* Complete brief assessments bi-weekly via phone for 1-year following treatment.
* Complete in-person interviews at 3 or 6-month intervals post-treatment.

DETAILED DESCRIPTION:
The aim of the current application is to examine the utility and validity of National Institute on Alcohol Abuse and Alcoholism's (NIAAA)new definition of recovery within the context of a novel theoretical model. The proposed study will recruit participants seeking treatment for Alcohol Use Disorder (AUD) from the community. Participants will complete a structured clinical interview and provide information on their current alcohol use and related behaviors. All participants will receive 12 weeks of AUD psychotherapy and complete brief assessments at the end of each treatment session and biweekly during the first 12-months post treatment. In addition, participants will complete in-person interviews at 3-month and 6-month intervals post-treatment for the duration of the study (for up to 24-54 months post treatment depending on time of enrollment). Findings from the proposed research have the potential to increase understanding of the dynamic nature of recovery and thereby improve clinical decision-making and generate future research. Specifically, our goal is to address the question of "Are the constructs of relapse, recurrence remission, or recovery useful heuristics for clinical practice and research, and if so, how?"

ELIGIBILITY:
Inclusion Criteria:

1. current diagnosis of AUD (initial screening AUDIT ≥ 8, confirmed with diagnostic interview),
2. live within commuting distance of the program site,
3. provide informed consent.

Exclusion Criteria:

1. acute psychosis or severe cognitive impairment (assessed via Psychotic Module of the M.I.N.I and Mini-Mental State ≤ 23),
2. current drug use diagnosis other than nicotine or marijuana use disorders,
3. lack of sufficient familiarity with the English language to comprehend the recruitment and consent procedures,
4. legally mandated to attend treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2023-05-09 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Heavy Drinking Days (Timeline Follow-back assessment) | Administered at several timepoints during the study - weekly during treatment (first 3-months), biweekly (1-year following treatment), 3- and 6-month intervals (through completion of study, average between 24-48 months depending on enrollment date)
  Change in self-report percentage of Heavy Drinking Days, completed during interview with a research assistant.
Short Inventory of Problems-Alcohol (SIP-A) | Administered at several timepoints during the study - weekly during treatment (first 3-months), biweekly (1-year following treatment), 3- and 6-month intervals (through completion of study, average between 24-48 months depending on enrollment date)
  Self-report questionnaire that will measure change in negative consequences (e.g., quality of work has suffered due to alcohol, physical health has been harmed due to drinking, family has been hurt due to drinking) associated with alcohol use. Scores range from 0-45, with higher numbers indicating greater negative consequences associated with alcohol use.
Alcohol Dependence Scale (ADS) | Administered at several timepoints during the study - weekly during treatment (first 3-months), biweekly (1-year following treatment), 3- and 6-month intervals (through completion of study, average between 24-48 months depending on enrollment date)
  Self-re[port questionnaire will be used to measure change in the severity of alcohol dependence (e.g., frequency of hangovers, presence of withdrawal symptoms) - Scores range from 0 to 47, with higher scores indicating greater alcohol dependence severity.

SECONDARY OUTCOMES:
World Health Organization Quality of Life Scale-BREF (WHOQOL-BREF) | Administered at several timepoints during the study - Baseline, End of Treatment, 3- and 6-month intervals (through completion of study, average between 24-48 months depending on enrollment date)
  Self-report questionnaire that assesses change in overall quality of life across several domains (e.g., physical, psychological, social, environmental). Scores ranging between 0-100, with higher scores indicating higher quality of life.
12-Item Short-Form Health Survey (SF-12) | Administered at several timepoints during the study - Baseline, End of Treatment, 3- and 6-month intervals (through completion of study, average between 24-48 months depending on enrollment date)
  Self-report questionnaire measuring change in overall physical and mental health. Scores range from 0-100, with higher scores indicating greater health related problems.

CONTACTS AND LOCATIONS:
Locations (1):
- University of South Florida, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
In compliance with the grant funding agency (NIH/NIAAA, NOT-AA-22-011), participants who give consent will have all their de-identified survey/questionnaire data submitted and shared within the NIAAA Data Archive, which is a data repository housed within the NIMH Data Archive (NDA).
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Per NIAAA data sharing policy, there will be a 2-year embargo on data uploaded to the archive (i.e., data will only be shared 2 years after the grant end date on the initial NOA).
Access Criteria: Researchers can request de-identified data stored on NIAAA's data archive via submission of a data access request. Researchers (and the institution to which they belong) who requests data must promise to keep data safe and promise not to try to learn the identity of individual study records. Researchers submitting Data Access Requests must be sponsored by an NIH recognized institution (with a FWA) and have a research-related need to access NDA data.
  Request includes an NDA Data Use Certification signed by the lead recipient and an authorized Signing Official from the recipient's research institution. Data Access Requests for a given NDA Permission Group are reviewed by an NIH-staffed Data Access Committee.